CLINICAL TRIAL: NCT06017791
Title: Management of Excess Gingival Display Using Tunnel Technique With 3D Designed PEEK Shell: A Case Series
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farah Mamdouh Abdelfatah Mohamed Sheeba, Principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21623
Record Dates: First submitted 2023-08-17; First posted 2023-08-30 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Excessive Gingival Display

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEK shell in the anterior maxilla inserted by tunnel technique (Experimental): use of a minimally invasive tunnel technique to fill the skeletal subnasal depression with a PEEK shell in patients with an exaggerated subnasal depression associated with lack of lip support and excessive lip translation
  Interventions: Other: tunnel technique with a 3D printed PEEK shell to fill the skeletal subnasal depression

INTERVENTIONS:
Other: tunnel technique with a 3D printed PEEK shell to fill the skeletal subnasal depression — The area will be anesthetized using infiltration technique with 1.5ml of anesthetic solution containing Articaine Hydrochloride 68 mg/1.7 ml with Adrenaline 0.017 mg/1.7 ml
  Two bilateral full thickness vertical incisions will be created using a #15 blade. One on each side of the frenum
  A subperiosteal tunnel connecting the two vertical incisions will be created using a periosteal elevator/tunneling knife until the complete communication between the two ends is established
  The custom made PEEK framework will be inserted from the incision on one side and eased through until it sits in the subnasal concavity.
  Once fitted in place the shell will be fixed in place using two mini screws bilaterally, one on each side.
  The two vertical incisions will be closed by interrupted sutures 6-0 Polyglycolic acid suture material

SUMMARY:
The aim of the current study is to evaluate the use of a PEEK shell placed in the anterior maxilla placed by tunnel technique in decreasing the gingival display

DETAILED DESCRIPTION:
While lip repositioning has been established as a treatment modality to address excess gum display (EGD) , an often overlooked contributing factor is the lack of lip support. This is often caused by the architecture of the maxilla at the subnasal area. Maxillary overgrowth may give rise to a subnasal skeletal depression producing decreased lip support and marked upper lip retraction during a smile.

Restricting muscle pull by lip repositioning surgery as a treatment option limits muscle movement, however it does not address lip support. In 2018 an alternative intervention was later proposed in a case report study . The technique involves raising a full thickness flap and applying PMMA (polymethyl methacrylate) cement to fill the subnasal depression and limit the upper lip movement. Since its introduction, a limited number of studies have attempted to investigate the technique, however there are not enough studies to support the outcome or the stability of the technique. The aim of the current study is to evaluate the use of a tunnel technique with a 3D printed PEEK (Polyetherether ketone) shell to fill the skeletal subnasal depression

ELIGIBILITY:
Inclusion Criteria:

* Patients with excess gingival display 2.5mm or more
* Patients with an exaggerated subnasal concavity
* Decreased/normal value of SNA ( angle between sella, nation, A point) in cephalometric measurement
* Decreased/normal cephalometric measurement of A to N-perpendicular (perpendicular from N on FHP)
* Decreased/normal value in cephalometric measurement of the convexity at point A (linear measurement from point A to facial plane)
* Decreased/normal value of Ricketts Esthetic plane in cephalometric measurement
* Decreased/normal value of Holdaway H-angle in cephalometric measurement
* Nasolabial angle range from 100° to 120°
* Patients 20-60 years old
* Medically free
* Compliant patient that agrees to the follow up period

Exclusion Criteria:

* Pregnant and lactating females
* Smokers
* Diabetics
* Patients with parafunctional habits that may affect the outcome of the procedure
* Medically compromised patients

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Gingival display | Day 0 - Month 3 - Month 6
  measured using a periodontal probe in millimeters

SECONDARY OUTCOMES:
lip translation | Day 0 - Month 3 - Month 6
  measured using a periodontal probe in millimeters
profile angle | Day 0 - Month 6
  lateral cephalometric xray
lip length | Day 0 - Month 3 - Month 6
  measured using a periodontal probe in millimeters
patient satisfaction | Day 7
  measured by a binary Questionnaire ( yes or no)
Post operative pain | Day 7
  Measured by the visual analogue scale ( 0 no pain, 10 worst pain)
blinded esthetic assessment | Month 3- Month 6
  measured by a binary scale (yes or no)

CONTACTS AND LOCATIONS:
Locations (1):
- Farah Mamdouh, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 2025

REFERENCES:
- [Background] Brizuela M, Ines D. Excessive Gingival Display. 2023 Mar 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470437/ PMID 29262052
- [Background] El-Bokle, Dalia & Ghany, Amany. (2022). A sequential diagnostic scheme for excessive gingival display (Gummy Smile). AJO-DO Clinical Companion. 2. 10.1016/j.xaor.2022.05.003
- [Background] Impellizzeri A, Palmigiani R, Horodynski M, D'alfonso T, Polimeni A, De Stefano A, Galluccio G. Is There a Correlation between Gingival Display and Incisal Inclination in a Gummy Smile? Study on Cephalometric Parameters. Healthcare (Basel). 2023 Jan 25;11(3):344. doi: 10.3390/healthcare11030344. PMID 36766919
- [Background] Monaco A, Streni O, Marci MC, Marzo G, Gatto R, Giannoni M. Gummy smile: clinical parameters useful for diagnosis and therapeutical approach. J Clin Pediatr Dent. 2004 Fall;29(1):19-25. doi: 10.17796/jcpd.29.1.y01l3r4m06q3k2x0. PMID 15554398
- [Background] Toth, J. M. (2012). Biocompatibility of Polyaryletheretherketone Polymers. PEEK Biomaterials Handbook, 81-92. doi:10.1016/b978-1-4377-4463-7.10007-7
- [Background] Freitas de Andrade P, Meza-Mauricio J, Kern R, Faveri M. Labial Repositioning Using Print Manufactured Polymethylmethacrylate- (PMMA-) Based Cement for Gummy Smile. Case Rep Dent. 2021 Dec 21;2021:7607522. doi: 10.1155/2021/7607522. eCollection 2021. PMID 34970460
- [Background] Labial repositioning using polymethylmethracylate (PMMA)-based cement for esthetic smile rehabilitation-A case report Toni Arcuri a, Maykson Feitosa Pereira da Costa b, Iury Machado Ribeiroa, Byron Daia Barreto Júnior b, João Paulo Lyra eSilvac,∗ a Department of Dentistry, Paulista University, UNIP, Brasília, Brazil b Private Office in Brasilia, Brazil c Department of Dentistry, Universitary Center Euro Americano, UNIEURO, Brasília, Brazil
- [Background] ASSENZA, B. & Carinci, Francesco & CRISTINZI, A. & Sinjari, Bruna & Murmura, Giovanna & Scarano, Antonio. (2011). A COSMETIC TECHNIQUE CALLED LIP REPOSITIONING IN PATIENT OF EXCESSIVE GINGIVAL DISPLAY. European Journal of Inflammation. 9. 115-119.
- [Background] Dym H, Pierre R 2nd. Diagnosis and Treatment Approaches to a "Gummy Smile". Dent Clin North Am. 2020 Apr;64(2):341-349. doi: 10.1016/j.cden.2019.12.003. Epub 2020 Jan 24. PMID 32111273
- [Background] Saleem R, Kukreja BJ, Goyal M, Kumar M. Treating short upper lip with "Unified lip repositioning" technique: Two case reports. J Indian Soc Periodontol. 2022 Jan-Feb;26(1):89-93. doi: 10.4103/jisp.jisp_90_20. Epub 2022 Jan 1. PMID 35136324